CLINICAL TRIAL: NCT02230488
Title: Intensive Case Diabetes Management to Prevent Readmission of Previously Identified High Risk Patients
Brief Title: Intensive Case Diabetes Management (ICDM) to Prevent Readmission
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll due to protocol exclusion criteria and participant population pool
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201405143
Record Dates: First submitted 2014-08-26; First posted 2014-09-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes
Keywords: Inpatient Diabetes Management; Prevent <31 day readmission in patients with Diabetes; CDEs role in transition of care of inpatients with diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Diabetes Case Management (Active Comparator): Intensive Case Diabetes Management : A diabetes team , led by an endocrinologist and CDE, will manage the patients diabetes while in the hospital and will assist with the patient's discharge Diabetes endocrine consult team will manage the patient's diabetes daily while in the hospital Discharge diabetes medication reconciliation per research team Research team will provide 30 day supply of diabetes medication/supplies at discharge Research Team will provide 30 day supply of glucose test strips at discharge Discharge telecommunication from endocrinologist to primary care provider Patient-centered discharge diabetes education per research CDE Post-discharge 48-72 hours continuity check per phone by a diabetes research team member/CDE
  Interventions: Other: Intensive Diabetes Case Management
- Control :Standard/ usual care (No Intervention)

INTERVENTIONS:
Other: Intensive Diabetes Case Management — A diabetes team , led by an endocrinologist and CDE, will manage the patients diabetes while in the hospital and will assist with the patient's discharge Diabetes endocrine consult team will manage the patient's diabetes daily while in the hospital Discharge diabetes medication reconciliation per research team Research team will provide 30 day supply of diabetes medication/supplies at discharge Research Team will provide 30 day supply of glucose test strips at discharge Discharge telecommunication from endocrinologist to primary care provider Patient-centered discharge diabetes education per research CDE Post-discharge 48-72 hours continuity check per phone by a diabetes research team member/CDE
  --------------------------------------------------------------------------------
  Arms: Intensive Diabetes Case Management

SUMMARY:
The purpose of this study is to assess whether intensive case management interventions by a diabetes team, led by an endocrinologist and certified diabetes educator, can prevent <31 day readmission in previously identified high risk patients with diabetes.The procedures of the study will focus on managing the patient's diabetes and diabetes education while in the hospital, decreasing the patient's risk for hypoglycemia and hyperglycemia in the hospital, and assist in the patient's diabetes management plan for a safe discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with a diagnosis of diabetes, Patients with a previous history of Pharmacy Expert System (PES) alert, Enrollment in research must be within 24 hours of admission

Exclusion Criteria:

* Patients transferred from institutionalized care, Patients who already plan to move to institutionalized care, Patients with severe co-morbidities (e.g. terminal cancer), Patients admitted for surgery within 24 hours, Patients who are unwilling or unable to give written consent (e.g. dementia), Patients who are homeless, Patients previously admitted to the diabetes endocrine service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Prevent <31 day readmission | The length of time between hospital discharge and readmission 31 days
  Primary outcome measure is to assess whether an intensive case management intervention by a diabetes team, led by an endocrinologist and a certified diabetes educator (CDE) , can prevent a <31 day readmission in previously identified high risk patients with diabetes compared to standard/usual care.

SECONDARY OUTCOMES:
improve overall glycemic management | Upon the participant's consent (within 24 hours of hospital admission) to hospital discharge- the average length of stay is five days
  To examine whether intensive case management intervention per endocrinologist and CDE during hospital stay prevents hypoglycemia <70mg/dl, severe hypoglycemia <40mg/dl, and improves overall glycemic management (100-180 mg/dl) compared to standard/usual care.

OTHER OUTCOMES:
Patient satisfaction | From the time of consent (within 24 hours of admission) to the time of discharge- the average length of stay is 5 days.
  to assess whether intensive case management intervention by a diabetes team , led by an endocrinologists and a CDE, can improve patient's overall satisfaction.
  The research participant will be given a brief satisfaction questionaire at the time of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Garry Tobin, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States